CLINICAL TRIAL: NCT07064759
Title: A Phase 3, Randomized, Double-Masked, Active-Controlled Trial of a Single Intravitreal Injection of 4D-150 in Adults With Macular Neovascularization Secondary to Age-Related Macular Degeneration
Brief Title: Single Intravitreal (IVT) Injection of 4D-150 in Patients With Macular Neovascularization Secondary to Age-Related Macular Degeneration
Acronym: 4FRONT-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: 4D Molecular Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4D-150-C004
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Neovascular Age-Related Macular Degeneration (nAMD)
Keywords: Age-related macular degeneration; AMD; Exudative AMD; Neovascular AMD; Exudative age-related macular degeneration; Neovascular age-related macular degeneration; Wet age-related macular degeneration; Wet macular degeneration; Wet AMD; WAMD; nAMD; Retinal gene therapy; Intravitreal gene therapy; Genetic Medicine; Ocular Gene Therapy; Gene Therapy; 4FRONT; 4FRONT-2
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration | interventions — aflibercept; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 4D-150 IVT (3E10 vg/eye) (Experimental)
  Interventions: Biological: 4D-150 IVT (3E10 vg/eye)
- Aflibercept (AFLB) 2 mg IVT (Active Comparator)
  Interventions: Biological: EYLEA® (aflibercept) Injection 2 mg (0.05mL)

INTERVENTIONS:
Biological: 4D-150 IVT (3E10 vg/eye) — If randomized to the 4D-150 treatment arm, 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1
  Arms: 4D-150 IVT (3E10 vg/eye)
Biological: EYLEA® (aflibercept) Injection 2 mg (0.05mL) — Eylea (aflibercept) will be administered at applicable visits
  Arms: Aflibercept (AFLB) 2 mg IVT

SUMMARY:
A Phase 3, Randomized, Double-Masked, Active-Controlled Trial in Adults with Macular Neovascularization Secondary to Age-Related Macular Degeneration

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years of age at time of consent
* MNV secondary to nAMD with IVT anti-VEGF treatment history in the study eye, defined as EITHER:

  1. Treatment naïve, i.e. no prior IVT anti-VEGF therapy OR
  2. Previously treated with no more than 4 IVT anti-VEGF injections due to nAMD and received diagnosis of nAMD no more than 6 months prior to the Screening Visit AND documented evidence of anatomical improvement and visual stability/improvement in response to previous IVT anti-VEGF treatment, as determined by the Investigator
* Active subfoveal MNV or juxtafoveal/ extrafoveal MNV with a subfoveal component (where activity is defined as evidence of SRF, IRF, subretinal hyperreflective material, or leakage) identified by fluorescein angiography (FA) or spectral domain optical coherence tomography (SD-OCT) , in the study eye, at the Screening Visit confirmed by the Reading Center
* Demonstrated clinical response to aflibercept and functional stability in the study eye as confirmed by the Reading Center
* BCVA between 25 and 78 ETDRS letters, inclusive (20/320-20/32 Snellen equivalent) in the study eye at the Screening Visit
* CST less than or equal to 500 microns in the study eye at screening visit, confirmed by the central reading center

Exclusion Criteria:

Ocular Conditions:

* MNV due to causes other than nAMD in either eye (Fibrosis, atrophy, or subretinal hemorrhage in the foveal central subfield (1 mm diameter)
* History of retinal detachment in the study eye
* History of or presence of active inflammation in either eye
* Glaucoma or intraocular hypertension requiring more than 2 topical medications for control

Ocular Treatments/Interventions:

* Any prior or concomitant treatment for MNV or vitreomacular-interface abnormalities, other than allowed prior IVT anti-VEGF in the study eye

Systemic Conditions and Considerations:

* Major illness or major surgical procedure in the 28 days prior to the Screening Visit
* Uncontrolled blood pressure
* Acute coronary syndrome, myocardial infarction or coronary artery revascularization, cerebrovascular accident, transient ischemic attack within 6 months of the Screening Visit
* History of autoimmune condition that may predispose to the development of uveitis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Best Corrected Visual Accuity (BCVA) Early Treatment for Diabetic Retinopathy (ETDRS) letter score at Week 52 | 52 Weeks

SECONDARY OUTCOMES:
Mean annualized number of aflibercept injections after Week 4 through Weeks 52 and 104 | 104 Weeks
Incidence and timing of aflibercept injections after Week 4 through Weeks 52 and 104 | 104 Weeks
Proportion of subjects not requiring aflibercept injections after Week 4 through Weeks 52 and 104 in the 4D-150 arm | 104 Weeks
Mean change from baseline in Central Subfield Thickness (CST) over time through Weeks 52 and 104 | 104 Weeks
Mean change from baseline in BCVA ETDRS letter score over time through Weeks 52 and 104 | 104 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julie Tsai, MD, Study Director — 4D Molecular Therapeutics
Locations (43):
- United States (25):
  - Barnet Dulaney Perkins Eye Center, Sun City, Arizona
  - Retina Associates, Tucson, Arizona
  - Retinal Diagnostic Center, Campbell, California
  - Retina Consultants of Orange County, Fullerton, California
  - West Coast Retina Medical Group, San Francisco, California
  - Southwest Retina Consultants, Durango, Colorado
  - ClearVista Clinical Research, Hudson, Florida
  - Retina Vitreous Associates of Florida, Tampa, Florida
  - Thomas Eye Group, Sandy Springs, Georgia
  - The Retina Care Center, Baltimore, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Mid Atlantic Retina Specialist, Hagerstown, Maryland
  - New York Presbyterian Hospital - Columbia University Medical Center, New York, New York
  - Vitreoretinal Consultants of NY, Westbury, New York
  - North Carolina Retina Associates, Cary, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Verum Research, LLC, Eugene, Oregon
  - Charleston Neuroscience Institute, LLC, Bluffton, South Carolina
  - Carolina Eyecare, Mt. Pleasant, South Carolina
  - Tennessee Retina, PC, Nashville, Tennessee
  - Southwest Retina Specialist - Panhandle Eye group, LLP, Amarillo, Texas
  - Texas Retina Associate, Dallas, Texas
  - Tyler Retina Consultants, Tyler, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Pacific Northwest Retina, Silverdale, Washington
- Charles Research Center, Buenos Aires, Argentina
- Zora Eye Hospital, Sofia, Bulgaria
- Internationale Innovative Ophthalmochirurgie GbR, Düsseldorf, Germany
- Hungary (5):
  - Budapest Retina Associates, Budapest
  - Semmelweis Egyetem - Szemészeti Klinika, Budapest
  - DE KK Ophthalmology Clinic, Debrecen
  - Ganglion Medical Center, Pécs
  - SzTE SZAKK Szemeszeti Klinika, Szeged
- Hayashi Eye Hospital, Fukuoka, Japan
- Latvia (2):
  - P.Stradins University Hospital, Riga
  - Riga East University hospital, Riga
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Aibili - Cec, Coimbra, Portugal
- Singapore (2):
  - Singapore Eye Research Institute (SERI), Singapore
  - Tan Tock Seng Hospital TTSH, Singapore
- Spain (2):
  - Clinica Bonanova de Cirugía Ocular, Barcelona
  - Hospital Universitario Virgen Macarena, Seville
- The Retina Clinic London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided, after deidentification, to qualified researchers with academic interest in AMD in compliance with ICMJE policy. Data or samples shared will be coded, with no Protected Health Information included. Additionally, descriptions of the study protocol, Statistical Analysis Plan (SAP), informed consent and clinical study report may be shared publicly. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party. Data requests can be submitted starting after final Clinical Study Report and the data will be made accessible for a duration determined by the Sponsor, and in accordance with ICMJE policy. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and SAP and execution of a Data Sharing Agreement (DSA).